CLINICAL TRIAL: NCT07300020
Title: Single-Dose Pharmacokinetics and Relative Bioavailability of a Novel Liquid Metformin Formulation (100 mg/mL and 250 mg/mL) Compared With Immediate-Release Metformin Tablets in Adult Subjects
Brief Title: PK and Relative Bioavailability of Novel Liquid Metformin vs Tablets
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aspargo Labs, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ASP-017-Met
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-Arm Crossover (Experimental)
  Interventions: Drug: Novel Liquid Metformin 100 mg/mL; Drug: Novel Liquid Metformin 250 mg/mL; Drug: Metformin Immediate-Release Tablet

INTERVENTIONS:
Drug: Novel Liquid Metformin 100 mg/mL — Single oral dose of a novel liquid metformin formulation at 100 mg/mL administered under fasting conditions in one treatment period.
Drug: Novel Liquid Metformin 250 mg/mL — Single oral dose of a novel liquid metformin formulation at 250 mg/mL administered under fasting conditions in one treatment period.
Drug: Metformin Immediate-Release Tablet — Single oral dose of standard immediate-release metformin tablet(s) administered under fasting conditions in one treatment period.

SUMMARY:
This is an open-label, randomized, three-period crossover study evaluating the single-dose pharmacokinetics and relative bioavailability of a novel liquid metformin formulation at concentrations of 100 mg/mL and 250 mg/mL compared with immediate-release metformin tablets in healthy adult subjects. All participants will receive each formulation in randomized sequence with washout periods between treatments. Serial blood samples will be collected to characterize metformin pharmacokinetic parameters, and safety and tolerability will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults 18 to 55 years of age, inclusive.

Body mass index (BMI) between 18.0 and 30.0 kg/m², inclusive.

Medically healthy based on medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory tests, in the opinion of the investigator.

Non-smoker or light smoker (10 or fewer cigarettes per day or equivalent) willing to abstain from smoking during confinement periods, as determined by the investigator.

Able to understand and provide written informed consent before any study-specific procedures are performed.

Willing and able to comply with all study requirements, including fasting requirements, visit schedules, and pharmacokinetic blood sampling.

Females of childbearing potential must use acceptable contraception as determined by the investigator.

Exclusion Criteria:

* Known hypersensitivity or contraindication to metformin or any component of the study formulations.

History or presence of any clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, neurologic, or psychiatric disease that, in the opinion of the investigator, could interfere with study participation or interpretation of results.

Estimated glomerular filtration rate (eGFR) less than 90 mL/min/1.73 m², or any clinically significant abnormality in clinical laboratory tests.

History of lactic acidosis.

Use of any prescription or over-the-counter medications, herbal products, or dietary supplements within 14 days before the first study dose, unless considered acceptable by the investigator.

Positive test for hepatitis B surface antigen, hepatitis C antibody, or HIV.

Positive urine drug screen or positive alcohol breath test at screening or at admission to the clinical unit.

Participation in another clinical trial or receipt of an investigational drug or device within 30 days or 5 half-lives of the prior investigational product (whichever is longer) before the first study dose.

Donation of 450 mL or more of blood, or significant blood loss, within 8 weeks before the first study dose.

Pregnant or breastfeeding females.

Women of childbearing potential not using acceptable methods of contraception.

Any condition or circumstance that, in the opinion of the investigator, would make the subject unsuitable for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve from Time Zero to Last Quantifiable Concentration (AUC₀-t) of Metformin | Up to approximately 24 to 36 hours postdose in each treatment period
Maximum Observed Plasma Concentration (Cmax) of Metformin | Up to approximately 24 to 36 hours postdose in each treatment period

IPD SHARING:
Plan to Share IPD: No